CLINICAL TRIAL: NCT02347085
Title: A Randomized, Phase IIIb, Two-period, Two-treatment Double-blind, Multi-center, Crossover Study to Evaluate the 24-hour Lung Function Profile in Subjects With Moderate to Very Severe COPD After 4 Weeks of Treatment With PT003 and Placebo MDI
Brief Title: 24-hour Lung Function in Subjects With Moderate to Very Severe COPD After Treatment With PT003 and Placebo MDI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: PT003012
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GFF MDI (PT003) (Experimental): Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI)
  Interventions: Drug: GFF MDI (PT003)
- Placebo MDI (Placebo Comparator): Placebo Metered Dose Inhaler (MDI) for Glycopyrronium and Formoterol Fumarate Inhalation Aerosol
  Interventions: Drug: Placebo MDI

INTERVENTIONS:
Drug: GFF MDI (PT003)
  Other Names: Glycopyrronium and Formoterol Fumarate Inhalation Aerosol; PT003, Glycopyrronium and Formoterol Fumarate Metered Dose Inhaler (GFF MDI)
  Arms: GFF MDI (PT003)
Drug: Placebo MDI
  Other Names: Placebo Metered Dose Inhaler (MDI) for Glycopyrronium and Formoterol Fumarate Inhalation Aerosol
  Arms: Placebo MDI

SUMMARY:
Randomized, Phase IIIb, Two-period, Two-treatment Double-blind, Multi-center, Crossover Study to Evaluate the 24-hour Lung Function Profile in Subjects with Moderate to Very Severe COPD after 4 Weeks of Treatment with PT003 and Placebo MDI

ELIGIBILITY:
Inclusion Criteria:

* At least 40 years of age and no older than 80 at Screening
* Women of non-child bearing potential or negative serum pregnancy test at Screening, and agrees to acceptable contraceptive methods used consistently and correctly Screening until 14 days after final visit
* Subjects with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS)
* Current or former smokers with a history of at least 10 pack-years of cigarette smoking
* Pre- and post-bronchodilator FEV1/FVC ratio of <0.70
* Post-bronchodilator FEV1 must be <80% predicted normal value, calculated using NHANES III reference equations, and the measured FEV1 must also be ≥750 mL if FEV1 <30% of predicted normal value

Exclusion Criteria:

* Significant diseases other than COPD, i.e., disease or condition which, in the opinion of the Investigator, may put the subject at risk because of participation in the study or may influence either the results of the study or the subject's ability to participate in the study
* Women who are pregnant or lactating
* Subjects, who in the opinion of the Investigator, have a current diagnosis of asthma
* Subjects who have been hospitalized due to poorly controlled COPD within 3 months prior to Screening or during the Screening Period
* Subjects who have poorly controlled COPD, defined as acute worsening of COPD that requires treatment with oral corticosteroids or antibiotics within 6 weeks prior to Screening or during the Screening Period
* Subjects who have clinically significant uncontrolled hypertension.
* Subjects who have cancer that has not been in complete remission for at least five years
* Subjects with abnormal liver function tests defined as AST, ALT, or total bilirubin ≥1.5 times upper limit of normal at Screening and on repeat testing
* Subjects with a diagnosis of angle closure glaucoma will be excluded, regardless of whether or not they have been treated. Subjects with a diagnosis of open angle glaucoma who have intraocular pressure controlled with medication(s) are eligible
* Subjects with symptomatic prostatic hypertrophy that is clinically significant in the opinion of the Investigator. Subjects with a trans-urethral resection of prostate (TURP) or full resection of the prostate within 6 months prior to Screening are excluded from the study
* Subjects with bladder neck obstruction or urinary retention that is clinically significant in the opinion of the Investigator

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, MD, Study Chair — Pearl Therapeutics

REFERENCES:
- [Derived] Reisner C, Gottschlich G, Fakih F, Koser A, Krainson J, Delacruz L, Arora S, Feldman G, Pudi K, Siddiqui S, Orevillo C, Maes A, St Rose E, Martin U. 24-h bronchodilation and inspiratory capacity improvements with glycopyrrolate/formoterol fumarate via co-suspension delivery technology in COPD. Respir Res. 2017 Aug 18;18(1):157. doi: 10.1186/s12931-017-0636-4. PMID 28821260
- See also: Redacted Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4137&filename=PT003012_Protocol_FINAL_31Dec14_Redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 5 sites in the US from March 2015 to Jun 2015. The study was anticipated to run for approximately 6 months but not to expected to exceed 9 months.The study period was 11 to 17 weeks for each subject.
Pre-assignment Details: Complete crossover study to assess the efficacy and safety of GFF MDI vs. Placebo MDI. Each subject received 28 days of study treatment in each assigned treatment, with a minimum 7 day washout period between each of the 2 periods. By-treatment sequence tabulations of the data were not pre-specified.
Groups:
- Overall Study: All subjects randomized
Period: Overall Study
Arm/Group | Overall Study
Started | 43
GFF MDI 14.4/9.6 µg | 40
Placebo MDI | 40
Completed | 33
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 1
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 1
Not completed — Protocol Criteria | 2

BASELINE CHARACTERISTICS:
Population: The MITT Population was a subset of the ITT Population including the subjects who received treatment and had post-treatment efficacy data from both treatment periods.
Arm/Group | All Subjects
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: FEV1 AUC0-24 on Day 29
Description: Forced Expiratory Volume in One Second (FEV1) Area Under the Curve (AUC)0-24 on Day 29
Time Frame: Day 29
Population: Modified-Intent-to-Treat (MITT) Population
Measure: Mean (95% Confidence Interval); unit: Liters
Groups:
- GFF MD (PT003): GFF MDI 14.4/9.6 µg
- Placebo: Placebo MDI
Arm/Group | GFF MD (PT003) | Placebo
Number analyzed (Participants) | 35 | 31
Liters | 0.166 [0.110 to 0.222] | -0.083 [-0.143 to -0.024]

2. Secondary Outcome: FEV1 AUC12-24 on Day 29
Description: FEV1 AUC12-24 on Day 29
Time Frame: Day 29
Population: MITT Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MD (PT003) | Placebo
Number analyzed (Participants) | 35 | 31
Liters | 0.115 [0.055 to 0.175] | -0.127 [-0.191 to -0.063]

3. Secondary Outcome: FEV1 AUC0-12 on Day 29
Description: FEV1 AUC0-12 on Day 29
Time Frame: Day 29
Population: MITT Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MD (PT003) | Placebo
Number analyzed (Participants) | 35 | 31
Liters | 0.216 [0.157 to 0.276] | -0.039 [-0.103 to 0.025]

4. Secondary Outcome: Peak Change From Baseline in FEV1 on Day 29
Description: Peak Change From Baseline in FEV1 following evening Dose on Day 29
Time Frame: Day 29
Population: MITT Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MD (PT003) | Placebo
Number analyzed (Participants) | 35 | 31
Liters | 0.344 [0.275 to 0.412] | 0.050 [-0.023 to 0.124]

5. Secondary Outcome: Peak Change From Baseline in FEV1 on Day 29
Description: Peak Change From Baseline in FEV1 following the morning dose on Day 29
Time Frame: Day 29
Population: MITT Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MD (PT003) | Placebo
Number analyzed (Participants) | 35 | 31
Liters | 0.410 [0.338 to 0.482] | 0.134 [0.058 to 0.209]

6. Secondary Outcome: Morning Pre-Dose Trough FEV1 on Day 29
Description: Morning Pre-Dose Trough FEV on Day 29
Time Frame: Day 29
Population: MITT Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MD (PT003) | Placebo
Number analyzed (Participants) | 35 | 32
Liters | 0.130 [0.086 to 0.173] | -0.012 [-0.058 to 0.033]

7. Secondary Outcome: Morning Pre-Dose Trough FEV1 on Day 30
Description: Morning Pre-Dose Trough FEV1 on Day 30
Time Frame: Day 30
Population: MITT Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MD (PT003) | Placebo
Number analyzed (Participants) | 35 | 31
Liters | 0.090 [0.032 to 0.148] | -0.064 [-0.124 to -0.003]

8. Secondary Outcome: Peak Change From Baseline in Inspiratory Capacity (IC) Following the Evening Dose on Day 29
Description: Peak Change from Baseline in Inspiratory Capacity (IC) following the evening dose on Day 29
Time Frame: Day 29
Population: MITT Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MD (PT003) | Placebo
Number analyzed (Participants) | 34 | 30
Liters | 0.486 [0.369 to 0.603] | 0.105 [-0.019 to 0.229]

9. Secondary Outcome: Peak Change From Baseline in IC Following the Morning Dose on Day 29
Description: Peak Change from Baseline in IC following the morning dose on Day 29
Time Frame: Day 29
Population: MITT Population
Measure: Mean (95% Confidence Interval); unit: Liters
Arm/Group | GFF MD (PT003) | Placebo
Number analyzed (Participants) | 35 | 31
Liters | 0.543 [0.448 to 0.639] | 0.208 [0.106 to 0.310]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed consent up to the follow-up phone call 7-14 days after last dose of study drug.
Description: The Safety Population was defined as all subjects who were randomized to treatment regardless and received at least one dose of study treatment. Serious adverse events collected from the time the subject signed consent up to 14 days following the last dose of study drug.
Groups:
- GFF MDI PT003: GFF MDI 14.4/9.6 µg
Arm/Group | GFF MDI PT003 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/40 | 1/40
Other Adverse Events (participants affected / at risk) | 1/40 | 6/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI PT003 (N=40) | Placebo (N=40)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GFF MDI PT003 (N=40) | Placebo (N=40)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Hypertenstion (Vascular disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent its opinions, or the opinions of the publication committee, if these differ with the proposed publication.